CLINICAL TRIAL: NCT07349368
Title: Effectiveness and Cost-effectiveness of Simultaneous Screening and Intervention for Antenatal Depression and Anxiety Symptoms From a Transdiagnostic Perspective: A Scale-up Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fangbiao Tao, Professor, Anhui Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170358
Record Dates: First submitted 2025-12-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Antenatal Depression; Antenatal Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care group (No Intervention): no additional intervention
- Stratified iCBT group (Experimental): Stratified iCBT(Internet-based Cognitive Behavioral Therapy) Intervention plus usual care
  Interventions: Behavioral: implementation group

INTERVENTIONS:
Behavioral: implementation group — 1. screening during pregnancy and 42 days postpartum
  2. Stratified iCBT Intervention, usual care Low-intensity: Mild cases (EPDS≥9/GAD-7≥5) received 11 animated video sessions adapted from WHO's Thinking Healthy Programme manual. High-intensity: Moderate-severe cases (EPDS≥12/GAD-7≥10) received low-intensity components and supplemental telehealth counseling.
  Arms: Stratified iCBT group

SUMMARY:
This scale-up study aimed to explore the effectiveness of simultaneous screening and intervention of antenatal depression and anxiety in preventing postpartum depression and anxiety and how scale-up might be successfully achieved. The age was ≥18 years old pregnancy and capable of completing the independent assessment of smart phones. Exclude those with abnormal comprehension and expression abilities. The implementation group, 1. screening during pregnancy and 42 days postpartum; 2. Stratified iCBT Intervention, usual care. Low-intensity: Mild cases (EPDS≥9/GAD-7≥5) received 11 animated video sessions adapted from WHO's Thinking Healthy Programme manual. High-intensity: Moderate-severe cases (EPDS≥12/GAD-7≥10) received low-intensity components and supplemental telehealth counseling. The control group, screening at 42 days postpartum, usual care.

ELIGIBILITY:
Inclusion Criteria:

* The age was ≥18 years old pregnancy and capable of completing the independent assessment of smart phones.

Exclusion Criteria:

* Exclude those with abnormal comprehension and expression abilities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3314 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) Score | at 42 days postpartum
  The EPDS is a 10-item self-report questionnaire. Total scores range from 0 to 30, with higher scores indicating more severe depressive symptoms.
Generalized Anxiety Disorder 7-item (GAD-7) Scale Score | at 42 days postpartum
  The GAD-7 is a 7-item self-report questionnaire. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.

OTHER OUTCOMES:
cost-effectiveness ratios (ICER) | at 42 days postpartum
  ICER were calculated by dividing the difference in mean costs by the difference in anxiety and/or depression symptoms-free (Δcosts/Δoutcome). Cost included screening, access to the animated videos, and counselling.

CONTACTS AND LOCATIONS:
Locations (1):
- Jieshou Maternal and Child Health Hospital, Fuyang, China

IPD SHARING:
Plan to Share IPD: No
This study does not currently plan to share individual participant data (IPD). The main reasons are: ① The study involves sensitive clinical information (e.g., scores from mental health scales), and there remains potential privacy risks even after de-identification; ② The data usage agreement does not include authorization for external sharing, and additional informed consent from study participants is required.